CLINICAL TRIAL: NCT05383079
Title: Combination of Radium-223 and Lutetium-177 PSMA-I&T in Men with Metastatic Castration-Resistant Prostate Cancer
Acronym: AlphaBet
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21/029
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2024-11

CONDITIONS: Metastatic Castration-resistant Prostate Cancer; MCRPC; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radium-223

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Radium-223 and Lutetium-177 PSMA-I&T (Experimental): In this single-arm study, patients will receive 7.4 GBq of 177Lu-PSMA-I&T on Day 1 of every 6 week Cycle. Radium-223 will be administered concurrently every 6 weeks. The dose of Radium-223 will vary in dose-escalation. Up to 6 Cycles will be given.
  Interventions: Drug: Lutetium-177 PSMA-I&T; Drug: Radium-223

INTERVENTIONS:
Drug: Lutetium-177 PSMA-I&T — Patients will be given 7.4 GBq of 177Lu-PSMA every 6 weeks for up to 6 Cycles
Drug: Radium-223 — During dose escalation, doses of Radium-223 that will be administered include 27.5 kBq/kg and 55 kBq/kg. The maximum tolerated dose of Radium-223 will be used during dose expansion. Radium-223 will be given once every 6 weeks for up to 6 doses between day 1-5 of each Cycle.

SUMMARY:
This clinical trial will evaluate the safety of Radium-223 in combination with 177Lu-PSMA-I&T in metastatic castration-resistant prostate cancer: Phase I/II study

DETAILED DESCRIPTION:
This prospective, single-centre, single-arm, open label, phase I/II trial will assess and establish the maximum tolerated dose (MTD), dose-limiting toxicities (DLTs), and recommended phase 2 dose (RP2D) of Radium-223 in combination with 177Lu-PSMA-I&T in patients with mCRPC.

36 men with mCRPC who have progressed on second-generation AR antagonist will be enrolled in this trial in two stages: dose escalation and a dose expansion phase over a period of 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be ≥ 18 years of age and must have provided written informed consent.
* Histologically or cytologically confirmed adenocarcinoma of the prostate, OR unequivocal diagnosis of metastatic prostate cancer. (i.e. involving bone or pelvic lymph nodes or para-aortic lymph nodes) with an elevated serum PSA.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
* Patients must have progressed on ≥ 1 second-generation AR-targeted agent (e.g., enzalutamide, abiraterone, apalutamide, or darolutamide).
* Patients must have progressive disease for study entry. PCWG3 defines this as any one of the following:

  * PSA progression: minimum of two rising PSA values from a baseline measurement with an interval of ≥ 1 week between each measurement.
  * Soft tissue progression as per RECIST 1.1 criteria
  * Bone progression: ≥ 2 new lesions on bone scan
  * Symptomatic progression eg. Bone pain
* At least three weeks since receiving anti-cancer treatment (other than ADT), the completion of surgery or radiotherapy prior to registration.
* Prior surgical orchiectomy or chemical castration maintained on luteinizing hormone-releasing hormone (LHRH) analogue (agonist or antagonist).
* Serum testosterone levels ≤ 1.75nmol/L (≤ 50ng/dL) within 28 days before registration.
* Significant PSMA avidity on PSMA PET/CT, defined as a minimum uptake of SUVmax 20 at a site of disease, and SUVmax >10 at sites of measurable disease >10mm (unless subject to factors explaining a lower uptake, e.g. respiratory motion, reconstruction artefact).
* ≥ 2 bone metastases must be present on bone scintigraphy which have not been previously treated with radiotherapy.
* No contraindication to treatment with a bone antiresorptive agent such as denosumab or zoledronic acid.
* Patients must have adequate bone marrow, hepatic and renal function documented within 28 days prior to registration, defined as:

  * Haemoglobin ≥ 90 g/L independent of transfusions (no red blood cell transfusion in last four weeks)
  * Absolute neutrophil count ≥ 1.5x10^9/L
  * Platelets ≥ 150 x10^9/L
  * Total bilirubin ≤ 1.5 x upper limit of normal (ULN) except for patients with known Gilbert's syndrome, where this applies for the unconjugated bilirubin component.
  * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 x ULN if there is no evidence of liver metastasis or ≤ 5 x ULN in the presence of liver metastases
  * Albumin ≥ 25 g/L
  * Adequate renal function: patients must have a creatinine clearance estimated of ≥ 40 mL/min using the Cockcroft Gault equation
* Sexually active patients are willing to use medically acceptable forms of barrier contraception.
* Willing to undergo biopsies, if disease is considered accessible and biopsy is feasible.
* Willing and able to comply with all study requirements, including all treatments and the timing and nature of all required assessments.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from study entry:

* Superscan on Bone scan (WBBS) or diffuse marrow involvement on PSMA PET/CT
* Prior treatment with 223Ra or 177Lu-PSMA.
* Has received more than one previous line of chemotherapy for the treatment of metastatic prostate cancer.
* Sites of discordant FDG-positive disease defined by minimal PSMA-expression and no uptake on WBBS (for bone metastases).
* Other malignancies within the previous 2 years other than basal cell or squamous cell carcinomas of skin or other cancers that are unlikely to recur within 24 months.
* Symptomatic brain metastases or leptomeningeal metastases.
* Patients with symptomatic or impending cord compression unless appropriately treated beforehand and clinically stable for ≥ four weeks.
* Concurrent illness, including severe infection that may jeopardise the ability of the patient to undergo the procedures outlined in this protocol with reasonable safety.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 36 (Estimated)
Dates: Start 2022-09-13 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting toxicities (DLTs) | Dose escalation phase is expected to be completed 6 months from the time the first patient is recruited.
  A DLT is defined as a toxicity that prevents further administration of the trial treatment at that dose level.
  Each cohort of 3 patients be assessed for DLTs in the first 6 weeks (cycle 1) of treatment and a dose for the next cohort will be determined.
Maximum Tolerated dose (MTD) | Dose escalation phase is expected to be completed 6 months from the time the first patient is recruited.
  The MTD is defined as the highest dose level at which the incidence of DLT was less than 2/6.
Recommended Phase 2 Dose (RP2D) | Up to 30 months from the time the first patient is recruited.
  After the MTD is established, additional patients will be treated at the MTD. Safety and efficacy data from the study will be used to define the RP2D.
50% Prostate-Specific Antigen Response Rate (PSA-RR) | Through study completion, up until 12 months after the last patient commences treatment
  PSA will be assessed at baseline and every 3 weeks from cycle 1 day 1. PSA response will be defined as a 50% or greater decrease in PSA from baseline to the lowest post-baseline PSA result. A second consecutive value obtained 3 or more weeks later is required to confirm the PSA response.

SECONDARY OUTCOMES:
Adverse Events and Serious Adverse Events measured using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0 | Through study completion, up until 12 months after the last patient commences treatment
  Safety of the combination will be measured by AEs and SAEs.
Radiographic Progression-Free Survival (rPFS) | Through study completion, up until 12 months after the last patient commences treatment
  rPFS is defined as the time from treatment initiation to the first date of documented radiographic progression using conventional imaging or death due to any cause, whichever occurs first. The radiographic progression will be assessed by the investigator per RECIST1.1 for soft tissue and PCWG3 for bone lesions.
PSA progression free survival (PSA-PFS) | Through study completion, up until 12 months after the last patient commences treatment
  PSA-PFS is defined as the time from treatment initiation to the date of PSA progression per PCWG3 or death due to any cause, whichever occurs first. The date of PSA progression is the date that an increase of 25% or more and an absolute increase of 2ng/mL or more from the nadir is documented. For patients who have an initial PSA decline during treatment, this must be confirmed by a second value 3 or more weeks later.
Overall survival (OS) | Through study completion, up until 12 months after the last patient commences treatment
  OS is defined as the time from treatment initiation to the date of death due to any cause.
Objective response rate (ORR) by RECIST1.1 in patients with measurable disease | Through study completion, up until 12 months after the last patient commences treatment
  Objective Response (OR) is only applicable for the subset of patients with measurable disease by RECIST1.1. OR is defined as a partial response (PR) or complete response (CR) at any stage from time of commencement of protocol treatment to the time of subsequent systemic anti-cancer treatment. The ORR is calculated as the proportion of patients with a best response of CR or PR.
Progression Free Survival (PFS) | Through study completion, up until 12 months after the last patient commences treatment
  Time from randomisation to the date of PSA progression, or radiographic progression (PCWG3 for bone and RECIST 1.1 for soft tissue), or death.
Describe pain within 12 months of treatment commencement | Through completion of 12 months after treatment commencement of last patient
  Pain will be assessed using the Brief Pain Inventory - Short Form (BPI-SF). The primary endpoint for pain is the area under the curve (AUC) of the worst pain in 24h.
  Pain and QoL will be assessed at baseline, 6 weeks, 3 months, 6 months, 9 months and 12 months and will be scored according to the respective manuals.
Describe health-related QoL within 12 months of treatment commencement | Through completion of 12 months after treatment commencement of last patient
  QoL will be assessed using the Functional Assessment of Cancer Therapy for Prostate Cancer (FACT-P) questionnaire. The primary endpoint for QoL is the area under the curve (AUC) of the trial outcome index (TOI).
  QoL will be assessed at baseline, 6 weeks, 3 months, 6 months, 9 months and 12 months and will be scored according to the respective manuals.

CONTACTS AND LOCATIONS:
Overall Officials: Prof Michael Hofman, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (1):
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kostos L, Buteau JP, Xie J, Cardin A, Akhurst T, Alipour R, Au L, Chan J, Chin KY, Emmerson B, Furic L, Garcia Q, Hamilton AJ, Haskali MB, Jackson PA, Kashyap RK, Kong G, MacFarlane L, Murphy DG, Parker BS, Ravi Kumar AS, Saghebi J, Wang Y, Tran B, Azad AA, Hofman MS. Lutetium-177 [177Lu]Lu-PSMA-I&T plus radium-223 in patients with metastatic castration-resistant prostate cancer (AlphaBet): an interim analysis of the investigator-initiated, single-centre, single-arm, phase 1/2 trial. Lancet Oncol. 2025 Nov;26(11):1479-1488. doi: 10.1016/S1470-2045(25)00559-5. Epub 2025 Oct 18. PMID 41119954
- [Derived] Kostos L, Buteau JP, Yeung T, Iulio JD, Xie J, Cardin A, Chin KY, Emmerson B, Owen KL, Parker BS, Fettke H, Furic L, Azad AA, Hofman MS. AlphaBet: Combination of Radium-223 and [17 7Lu]Lu-PSMA-I&T in men with metastatic castration-resistant prostate cancer (clinical trial protocol). Front Med (Lausanne). 2022 Nov 18;9:1059122. doi: 10.3389/fmed.2022.1059122. eCollection 2022. PMID 36465905